CLINICAL TRIAL: NCT00535912
Title: A Multicentric Phase III Study in Patients With CLL B and C < 60 Years Not Treated: 6 Montly CHOP + 6 CHOP Every 3 Months Versus 3 Montly CHOP + Intensification and Autograft
Brief Title: Phase III Study Treatment of CLL B and C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LLC 98
Record Dates: First submitted 2007-09-26; First posted 2007-09-27 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-09

CONDITIONS: Leukemia, Lymphocytic, Chronic
Keywords: CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (No Intervention): ¨Chemotherapy by 12 courses of CHOP
- B (Active Comparator): ¨Chemotherapy by 3 courses of CHOP, intensification and autograft
  Interventions: Procedure: Stem cells autograft

INTERVENTIONS:
Procedure: Stem cells autograft — Treatment by Intensive Chemotherapy and autograft
  Arms: B

SUMMARY:
GOELAMS LLC98 is a prospective randomized trial comparing in previously untreated B and C Binet stages B-CLL and on an intent to treat basis two strategies. Conventional chemotherapy consisted of six monthly courses of CHOP, followed by 6 CHOP courses every other 3 months in case of response. Experimental arm consisted of high dose therapy with autologous CD34+ purified progenitor cell support, used as consolidation of Complete Remission or Very Good Partial Response obtained after 3 monthly courses of CHOP, followed by 3 to 6 monthly-courses of fludarabine in case of insufficient response.

DETAILED DESCRIPTION:
The aim of the prospective randomized GOELAMS LLC 98 trial reported here was to compare two therapeutic strategies in previously untreated B and C Binet stages B-CLL patients less than 60 years old. Conventional chemotherapy (Arm A) consisted of six monthly courses of CHOP, i.e. vincristin IV 1 mg/m2 on day 1, doxorubicin IV 25 mg/m2 on day 1, cyclophosphamide (Cy) 300 mg/m2 and prednisone 40 mg/m2 both given orally from day 1 to day 5, followed by 6 CHOP courses every other 3 months in case of response. Fludarabine (25 mg/m2 /d IV for 5 consecutive days) was used in case of non response (stable disease or progression) after 3 CHOP courses. This conventional therapy was compared to high dose therapy with autologous CD34+ purified progenitor cell support (Arm B), used as consolidation of Complete Remission (CR) or Very Good Partial Response (VGPR, defined by >50 % tumoral response and bone marrow lymphocyte infiltration <30%) obtained after 3 monthly courses of CHOP. In the absence of CR or VGPR, 3 to 6 monthly-courses of fludarabine were performed before mobilization with Cy 4 g/m2 + G-CSF administration. The conditioning regimen included TBI 12 Gy and Cy 60 mg /kg /d for 2 days.

ELIGIBILITY:
Inclusion Criteria:

* CLL with Lymphocitis > 15.10 9/L
* B-CLL stage B or C
* Patients > 18 years old and < 60 years old
* No previous treatment of CLL
* ECOG performance status < 2
* Good cardiac function
* Patient's written informed consent

Exclusion Criteria:

* B-CLL stage A
* Age > 60 years old
* previous treatment of CLL
* ECOG performance status > 2
* Cardiac or pneumo Insufficency
* hepatic or renal Insufficency
* Seropositivity HIV
* Previous other malignancy
* Fertile male and female patients who cannot or do not wish to use an effective method of contraception
* Any coexisting medical or psychological condition that would preclude participation to the required study procedures
* NOt signed Patient's informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 1999-01; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
progression free survival | Overal survival

SECONDARY OUTCOMES:
response belong NIC criterias | 3 years after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Annie BRION, RN, Principal Investigator — French Innovative Leukemia Organisation